CLINICAL TRIAL: NCT05644197
Title: Effect of Psychological, Nutritional and Activity Support Physical on Recovery After Treatment by Prostatectomy for Localized Prostate Cancer
Brief Title: Multidisciplinary Care After Prostatectomy
Acronym: MCAP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Provence Private hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2021-A03118-33
Record Dates: First submitted 2021-12-16; First posted 2022-12-09 (Actual); Last update posted 2022-12-09 (Actual); Status verified 2022-11

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Intervention Model Description: the two groups will be followed in parallel, intervention group composed of 50 patients and control group composed of 50 patients, the duration of participation for each patient is 15 months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Other): the intervention group of 50 patients will undergo a support program over 12 weeks (1 adapted physical activity session per week, will participate in 5 workshops with the psychologist and 1 workshop with the dietician, plus a visit with the urologist after 6 weeks from prostatectomy
  Interventions: Other: Multidisciplinary program
- control group (No Intervention): the control group will only undergo a classic follow-up during its 12 weeks, namely a visit to the urologist after 6 weeks of the prostatectomy

INTERVENTIONS:
Other: Multidisciplinary program — Multidisciplinary program:
  * APA interventions: 12 weeks Each week at home, cardio-respiratory endurance sessions for muscle strengthening and balance work from the Autohome interface (Neuradom) and one week supervised by an APA teacher.
  * Nutrition interventions: A group nutrition workshop at the Hôpital Privé de Provence.
  * Psychological intervention:
    5 sessions of 1h30 in group, the first session will take place at the Private Hospital of Provence and the others by videoconference.
  An individual session the week following the last group session.
  -Visit with the urologist, 5 weeks after the prostatectomy.
  Arms: intervention group

SUMMARY:
This is a pilot, prostective, comparative, randomized, monocentric open-label study whose main objective is to determine whether appropriate psychological, nutritional and physical activity support can improve the quality of life of carrier patients. localized prostate cancer treated by prostatectomy

DETAILED DESCRIPTION:
Pilot study to demonstrate the benefits of a multimodal intervention (psychological and nutritional support and physical activity) on the recovery of patients treated by prostatectomy for localized prostate cancer.

After inclusion of 100 patients, at week 6 will undergo a prostatectomy and then at week 9 will be randomized into two groups of 50 patients for each group.

Groupe Intervention which will benefit from multidisciplinary care over 12 weeks (one APA session per week plus 5 workshops with the psychologist and a workshop with the dietician) plus a visit with the urologist.

Then after 3 months, 6 months and 12 months, the group benefit from an evaluation with the urologist, the teacher of adapted physical activity and the dietitian.

-For the control group, it will be followed classically, a visit to the urologist, an assessment with the teacher of physical activity and the dietician, after prostatectomy, then at 3 months, 6 months and at 12 months.

ELIGIBILITY:
Inclusion Criteria:

WHO score 0 or 1

* Adult patients with localized prostate cancer eligible for surgical treatment according to the AFU criteria following the CAPRA and d'Amico classifications: low risk or risk intermediaries. These are patients under the age of 73, with clinical stage and or MRI < or = T3, PSA < or = 20 ng/ml, with assessment negative extension (bone scintigraphy, thoraco-abdomino-pelvic scanner, Choline Pet-scanner)
* Informed and written consent signed by the patient
* Person affiliated with social security or beneficiary of such a scheme

Exclusion Criteria:

WHO score greater than or equal to 2

* MMSE score below 20
* Persons referred to in Articles L1121-5 to L1121-8 of the CSP (corresponds to all protected persons: person deprived of liberty by judicial or administrative decision, person subject to a legal protective measure)

Ages: 18 Years to 72 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-01 (Estimated); Primary Completion 2024-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Comparison of changes (over time) in quality of life for control and study groups | At baseline, 3 weeks after prostatectomy, 3, 6 and 12 months after start of intervention
  The program will focus on changes in quality of life. Quality of life will be measured using a questionnaire. Comparaison of changes in quality of life for control and study groups:
  Between patients treated with prostatectomy receiving either a standard or a multimodal therapy. At several time points during the study period, from baseline assessments(T0) up to follow up:3,6 and 12 months after start of intervention, using the Functional Assessments of Cancer Therapy-Prostate (FACT-P) questionnaire. With higher score correlating with better quality of life.
  Adapted Physics) at 3, 6, and 12 months will be studied using a model linear mixed

SECONDARY OUTCOMES:
Cardiorespiratory fitness assessment | From baseline assessments up to 3 weeks after prostatectomy
  Changes in cardiorespiratory fitness for all patients from baseline assessments up to 3 weeks after prostatectomy assessed either by the Luc Léger's Shuttle test or TM6, depending on the patient conditions. (m.s-1, /m.s)
Physical performance (quadriceps and biceps endurance tests) | From baseline assessments up to 3 weeks after surgery
  Changes in quadriceps and biceps strength for each individual patient from baseline assessments up to 3 weeks after surgery assessed by 2 items comprising the senior fitness test:- Quadriceps endurance test: The 30-Second Chair Stand or Sit to Stand Test/item for measuring lower body strength (Number of full stands that can be completed in 30 seconds with arms crossed at the wrists and held against the chest).
  -Biceps endurance test: The Arm Curl item for measuring upper body strength (Number of bicep curls that can be completed in 30 seconds holding a hand weight of 7.7 (3.5 kg), one arm at a time.
Emotional regulation assessment | 3 weeks after prostatectomy up to follow up: 3, 6 and 12 months after start of intervention
  Changes in emotion regulation strategies for each individual patient 3 weeks after prostatectomy up to follow up: 3 ,6 and 12 months after start of intervention using the cognitive emotional regulation questionnaire (CERQ).
  Higer score indicating greater difficulty in emotion regulation.
Anxiety assessment-Self reported anxiety level | From 3 weeks after prostatectomy up to follow up: 3, 6 and 12 months after start of intervention
  Changes in anxiety level for each individual patient from 3 weeks after prostatectomy up to follow up: 3, 6 and 12 months after start of intervention using the State Trait Inventory (STAI Y1 and Y2). Patients will be asked to score a series of questions split into the S-Anxiety scale that requires the participants to describe how they feel at this moment, and the T-Anxiety scale to describe how they generally feel, on a 4-pointscale. With higher scores indicating greater anxiety.
Well-being assessment | From 3 weeks after prostatectomy up to follow up: 3, 6 and 12 months after start of intervention
  Changes in psychological well-being (change in scores) for each individual patient from 3 weeks after prostatectomy up to follow up: 3,6 and 12 months after start of intervention using the Ryff Scales of Psychological Welle-being.
  Patients will be asked to rate how strongly they agree or disagree with 18 statements in 6 areas (autonomy, Environnemental Mastery, Personal Growth, Positive Relations with Others, Purpose in life, Self-acceptance) using a 6- point scale (1 = strongly agree; 6 = strongly disagree) with higher score indicating a better outcome.
Psychological distress (in terms of depression and anxiety) assessment | From 3 weeks after prostatectomy up to follow up:3, 6 and 12 months after start of intervention
  Changes in anxiety and/or depression symptoms (change in scores) for each individual patient from 3 weeks after prostatectomy up to follow up: 3, 6 and 12 months after start of intervention using the Hospital Anxiety and Depression Scale (HADS). Higher score indicating greater levels of anxiety or depression
Nutritional assessment/Nutrition-related variables | After prostatectomy up to follow up
  Changes in nutritional parameters for each individual patient after prostatectomy up to up follow up using the Subjective Global Assessment (SGA)
  * the acquisition of knowledge of the people treated with regard to food and its daily management as well as their behavior when using the tools (the different food groups, their roles, consumption benchmarks, knowledge of foods rich in energy, foods rich in protein...) by means of questionnaires.
  * improvement of nutritional status parameters
Patient adherence to nutritional care and support | From 3 weeks after prostatectomy up to 3 months after start of intervention and in the empowerment process at 6 and 12 months
  Patient adherence level during the supportive care intervention phase from 3 weeks after prostatectomy up to 3 months after start of intervention and in the empowerment process at 6 and 12 months, using the Subjective Global Assessment (SGA)
Assessing physical performance | After surgery up to follow up: at 3, 6 and 12 months
  Changes in physical performance for each individual patient after surgery up to follow up: at 3, 6 and 12 month using the Luc Léger's Shuttle test or TM6.
The quality of physical activity | At baseline, 3 weeks after prostatectomy, 3, 6 and 12 months after start of intervention
  The quality of physical activity during the program will be assessed for each individual patient from baseline assessments up to 3 weeks after prostatectomy up to follow up:3, 6 and 12 months after start of intervention using the International Physical Activity questionnaire. Patients will be asked to score a series of questions (frequency =number of days per week; duration (in minutes)) in 3 specific types of activities (Walking, moderate-intensity and vigorous-intensity activities). Undertaken in 4 domains (leisure time physical activity; domestic and gardening (yard) activities; work-related physical activity; transport-related physical activity). With higher score correlation with higher levels of physical activity
Physical Activity commitment | Patient adherence will be measured each month during the entire study.
  Patient engagement/adherence as a measure of Physical Activity commitment. Patient adherence will be measured each month during the entire study period 1) using Heart Rate Monitors/real-time heart rate feedback, 2) measuring daily energy expenditure, 3) comparing the number of sessions and duration of exercise par week with the recommended amount of weekly activity and 4) assessing session perceived exertion using the visual analog scale (vas)

CONTACTS AND LOCATIONS:
Overall Officials: Eve NEGRE, Psychologist, Study Chair — Provence Private hospital; Thibault NEGRE, Urologist, Study Chair — Provence Private hospital